CLINICAL TRIAL: NCT07094087
Title: A Phase 3, Multicenter, Randomized, Open-label, Controlled Study to Investigate the Efficacy and Safety of 4-Factor Prothrombin Complex Concentrate in Adult Patients Undergoing Complex Cardiovascular Surgery With Cardiopulmonary Bypass
Brief Title: Efficacy and Safety of 4F-PCC (4-Factor Prothrombin Complex Concentrate) in Adult Patients Undergoing Complex Cardiovascular Surgery With Cardiopulmonary Bypass (CPB)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BE1116_3008
Record Dates: First submitted 2025-07-14; First posted 2025-07-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Complex Cardiovascular Surgery With Cardiopulmonary Bypass
Keywords: Cardiopulmonary bypass; Coagulopathic Bleeding; Coagulation factor deficiency; Prothrombin complex concentrates; Fresh frozen plasma
MeSH Terms: interventions — Factor IX

STUDY DESIGN:
Intervention Model Description: This is multicenter, randomized, open-label, parallel group, controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BE1116 (Experimental)
  Interventions: Biological: BE1116
- Fresh frozen plasma (Active Comparator)
  Interventions: Biological: FFP

INTERVENTIONS:
Biological: BE1116 — A single dose of BE1116 will be administered by intravenous (IV) infusion intraoperatively.
  Other Names: 4F-PCC
  Arms: BE1116
Biological: FFP — A single dose of FFP will be administered as investigational product (IP) by IV infusion intraoperatively.
  Arms: Fresh frozen plasma

SUMMARY:
This is a phase 3, multicenter, randomized, open-label, parallel-group, controlled study to assess the efficacy and safety of BE1116 compared with fresh frozen plasma (FFP) in adult participants undergoing complex cardiovascular surgery with CPB. The primary purpose of the study is to compare the efficacy of BE1116 and FFP in correcting coagulation factor deficiencies in bleeding participants undergoing complex cardiovascular surgery with CPB.

ELIGIBILITY:
Inclusion Criteria:

* Adult greater than or equal to (≥) 18 years and has provided written informed consent.
* Undergoing elective complex cardiovascular surgery requiring CPB, including procedures of the thoracic aorta (with or without additional cardiac interventions), aortic valve replacement + coronary artery bypass graft (CABG), complex valve surgeries, mitral valve repair + CABG, and mitral valve replacement + CABG and reoperative CABG. Reoperative procedures are permitted. Excluded surgeries are as follows: heart transplantation, insertion or removal of ventricular assist devices (except for intra-aortic balloon pumps), and acute repair of thoracoabdominal aneurysms.
* Coagulation factor replacement (ie, 4F-PCC or FFP) is ordered in the operating room for the management of bleeding, in accordance with accepted clinical standards. The following criteria must be met:
* INR ≥ 1.6 (point-of-care INR testing by Hemochron ≥ 5 to 10 minutes after protamine infusion for heparin reversal). If a participant needs a second dose of protamine, a new INR measurement should be performed to confirm eligibility.
* Significant microvascular hemorrhage (ie, not due to surgical complications), as defined by a BSS score of ≥ 2.

Exclusion Criteria:

* Administration of any systemic hemostatic therapy, such as cryoprecipitate, platelets, FFP, PCC (eg, 4-factor / 3-factor PCC [4F-PCC / 3F-PCC]), Factor VIII (FVIII) inhibitor bypassing activity (FEIBA), recombinant activated Factor VIIa (rFVIIa), or other coagulation factor products, in the 24 hours before study surgery, except when FFP is added to the CPB circuit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-11-18 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With and Without a Successful Correction of Coagulation Factor Deficiency | At Day 1 after IP infusion (30 minutes after the end of infusion)
  Successful correction ("yes" vs "no") of coagulation factor deficiency as measured by an international normalized ratio (INR) of less than or equal to (≤) 1.4 at 30 minutes after the end of IP infusion.

SECONDARY OUTCOMES:
Number of Participants With Effective or Not Effective Hemostatic Response from 30 Minutes to 24 Hours After the End of IP Infusion | Up to 24 hours after the end of IP infusion
  The hemostatic response will be recorded as either effective or not effective. 'Effective' is defined as no hemostatic intervention was required, whereas 'non effective' is defined as a hemostatic intervention was required in the period from 30 minutes to 24 hours after the end of IP infusion. Hemostatic intervention includes surgical re-intervention for bleeding and / or the administration of any systemic hemostatic agents.
Number of Participants With and Without Successful Correction of Coagulation Factor Deficiency | At Day 1 after IP infusion (30 minutes after the end of infusion)
  Successful correction ("Yes or No") of coagulation factor deficiency measured by a rotational thromboelastometry (ROTEM) extrinsically activated thromboelastometric test (EXTEM) clotting time (CT) ≤ 80 seconds or thromboelastography (TEG) reaction time ≤ 8 minutes. ROTEM and TEG are viscoelastic coagulation tests that quantify the process of clot formation and degradation.
Change in INR from Baseline | From baseline (before IP infusion), to 30 minutes, 6 hours, 24 hours, and 48 hours after the end IP infusion
Number of Participants With Effective and Not Effective Hemostatic Response From the Start of IP Infusion to 24 Hours After the Start of IP Infusion | Up to 24 hours after the start of IP infusion
  The hemostatic response will be recorded as either effective or not effective. 'Effective' is defined as no hemostatic intervention was required, whereas 'non effective' is defined as a hemostatic intervention was required in the period from the start of IP infusion to 24 hours after the start of IP infusion. Hemostatic intervention includes surgical re-intervention for bleeding and / or the administration of any systemic hemostatic agents.
Change in Z-Scores for ROTEM EXTEM CT and TEG Reaction Time | From baseline (before IP infusion) to 30 minutes and 24 hours after the end IP infusion
  Measurements on either ROTEM EXTEM CT or TEG reaction time will be collected. To combine these measurements, z-scores will be calculated for each method of measurement. The z-score standardizes each measurement by subtracting the mean and dividing by the standard deviation of the respective method.
Change in Bleeding Severity Scale (BSS) Score From Baseline | From baseline (before IP infusion) to 30 minutes after end of IP infusion
  The BSS is a validated intraoperative scale used in clinical studies of hemostatic agents as a measure of bleeding severity. Bleeding is scored on a scale from 0 (no bleeding) to 4 (unidentified or inaccessible spurting or gush). A lower score indicates a better outcome.
Number of Participants in Each Universal Definition for Perioperative Bleeding (UDPB) Class | During surgery (Day 1) and on the first postoperative day (Day 2)
  Bleeding is assessed based on 9 events occurring during surgery or within the first postoperative day. These 9 events will be used to determine UDPB class ranging from Class 0 to 5 as follows: Class 0 (insignificant), Class 1 (mild), Class 2 (moderate), Class 3 (severe), and Class 4 (massive).
Total Number of Units of Allogeneic Blood Products (ABPs) Administered | From the start of IP infusion and up to 24 hours and 5 days after surgery
  The ABPs include whole blood, cryoprecipitate, platelets, red blood cells (RBCs), and FFP (except the dose administered as IP). For the purposes of this study, a dose of fibrinogen concentrate will be counted as an ABP, because it is administered in lieu of cryoprecipitate.
Number of Units of Individual ABPs Administered | Up to 24 hours after the start of IP infusion
  The ABPs include whole blood, cryoprecipitate, platelets, RBCs, and FFP (except the dose administered as IP). For the purposes of this study, a dose of fibrinogen concentrate will be counted as an ABP, because it is administered in lieu of cryoprecipitate.
Volume of Chest Tube Output | Up to 24 hours after the end of surgery
Number of Participants Requiring Reoperation for Bleeding and for Other Reasons | Up to 30 days after surgery
Duration of Mechanical Ventilation | Up to 30 days after surgery
  The duration of mechanical ventilation is defined as the number of days on mechanical ventilation after the study surgery. If there are multiple incidences of mechanical ventilation, the duration will be the sum of the number of days for all incidences.
Duration of Primary Intensive Care Unit (ICU) Stay | Up to 30 days after surgery
  The duration of primary ICU stay is defined as the number of days in the ICU after the study surgery.
Duration of Primary Hospital Stay | Up to 30 days after surgery
  The duration of primary hospital stay is defined as the duration in calendar days from the date of IP administration to the date of primary hospital discharge, or death in the hospital, or end of study (EOS) visit, whichever occurs first.
Number of Deaths | Up to Day 1 during the primary hospital stay, and within 28 days following IP infusion
Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, and Adverse Events of Special Interest (AESIs) | Up to 30 days after IP infusion
Change in Plasma Concentrations of Coagulation Factor II (FII), Factor VII (FVII), Factor IX (FIX), and Factor X (FX), and Proteins C and S From Baseline | From baseline to 30 minutes after the end of IP infusion
Plasma Concentrations of Coagulation FII, FVII, FIX, and FX and Proteins C and S | Up to 48 hours after the end of IP infusion

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- 84000877- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.